CLINICAL TRIAL: NCT05819229
Title: Oral Antibiotics Alone in Children Aged 4 Weeks to 2 Months With a Suspected or Confirmed Uncomplicated Urinary Tract Infection. A Single-arm Multicenter Prospective Observational Study.
Brief Title: Oral Antibiotics Alone in Children Aged 4 Weeks to 2 Months With a Urinary Tract Infection
Status: Recruiting | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Ulrikka Nygaard, Principal investigator, Rigshospitalet, Denmark
Other Study IDs: PO AB UTI
Record Dates: First submitted 2023-02-22; First posted 2023-04-19 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Urinary Tract Infections in Children
Keywords: Antibiotic therapy; Urinary tract infection; Children
MeSH Terms: conditions — Urinary Tract Infections | interventions — Anti-Infective Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Oral antibiotic therapy: Clinically stable (see eligibility criteria) children without any past high-risk medical history (see eligibility criteria) will initiate oral antibiotic therapy.
  Interventions: Drug: Oral antibiotic therapy

INTERVENTIONS:
Drug: Oral antibiotic therapy — Empirical choice: amoxicillin-clavulanic acid 50 mg/kg/day divided into three doses.
  If the sensitivity pattern is available, another oral antibiotic, preferably smaller-spectrum, can be used instead.
  Total duration of antibiotic therapy will be 10 days.

SUMMARY:
The goal of this prospective study is to investigate whether oral antibiotic therapy alone is feasible and safe in clinically stable children aged 4 weeks to 2 months without any past high-risk medical history with a suspected or confirmed urinary tract infection.

DETAILED DESCRIPTION:
All children aged 4 weeks to 2 months with a suspected urinary tract infection will be observed and examined by physicians and nurses as recommended by current guidelines. Children needing empirical antibiotic therapy will be admitted. The remaining will be contacted by phone if the urine culture is positive, and antibiotic therapy will be initiated if a urinary tract infection is still suspected due to persistent symptoms.

Clinically stable (see eligibility criteria) children without any past high-risk medical history (see eligibility criteria) will initiate oral antibiotic therapy. As empirical oral therapy, amoxicillin-clavulanic acid 50 mg/kg/day divided into 3 doses will be used. If the sensitivity pattern is available, a smaller-spectrum antibiotic can be used instead. If these children at any time point become clinically unstable or have a positive blood culture without suspected contamination, parenteral antibiotic therapy will be initiated. As empirical parenteral therapy, gentamicin 5 mg/kg once daily and ampicillin 100 mg/kg/day divided into 3 doses will be used. If the sensitivity pattern is available, another parenteral antibiotic regime can be used instead.

Admitted children can be sent home when they have clinically improved (judged by the physician) and have been hospitalized at least until the ward round the following day. Parents will be informed to contact the pediatric emergency department immediately if the child worsens or does not tolerate the antibiotics.

A physical or virtual follow-up will be conducted on day 3 (approximately 72 hours after treatment initiation) to ensure clinical improvement and treatment adherence. If needed, antibiotic therapy will be changed according to the sensitivity pattern. Children with a negative urine culture will be informed to stop antibiotic therapy.

The duration of antibiotic therapy will be 10 days. All children will undergo a renal ultrasound within the treatment period.

The above recommendations has been implemented as routine care. Hence, no parental consent is needed.

ELIGIBILITY:
INCLUSION CRITERIA:

1. Clinical suspicion of urinary tract infection irrespective of the presence of fever.
2. Clinically stable (i.e., not respiratory or circulatory affected, septic, or meningeal).
3. 4 weeks to 2 months of age (corrected age, if premature).

All children who do not receive any empirical antibiotic therapy but have a positive urine culture can be included if the clinical suspicion of urinary tract infection persists.

A positive urine culture is defined as:

* Suprapubic bladder aspiration: any growth of bacteria.
* Sterile intermittent catheterization: monoculture with ≥10^3 colony forming units per milliliter (cfu/ml).
* Midstream urine x 2: monoculture with the same bacteria in both tests with ≥10^4 cfu/ml.
* Midstream urine x 2: monoculture with the same bacteria in both tests with ≥10^5 cfu/ml in one test and 10^3 cfu/ml in another test.

EXCLUSION CRITERIA:

1. Non-Danish civil registration number.
2. High-risk medical history.

   1. Previous urinary tract infection.
   2. Prophylactic antibiotic treatment.
   3. Known urogenital abnormality (i.e., hydronephrosis (pyelectasis ≥10 mm or/and caliectasis ≥5 mm); hydroureter; vesicoureteral reflux; multicystic dysplasia; renal dysplasia; renal hypoplasia; renal agenesis; duplex kidney; ectopic placed kidneys; polycystic kidney disease; neurogenic bladder dysfunction; and hypospadias).
   4. Previous hospitalization needing antibiotic therapy.
3. Markedly elevated c-reactive protein indicating bacteremia.
4. Elevated creatinine.
5. Oral therapy is not possible (e.g., frequent vomiting or excessive regurgitation).

Ages: 4 Weeks to 2 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All children aged 4 weeks to 2 months who are referred by their primary physician or the medical helpline 1813 (outside the work hours of their primary physician) to one of four pediatric emergency departments in the Capital Region of Denmark with suspected urinary tract infection.
Sampling Method: Non-Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2023-02-27 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with recurrent urinary tract infection regardless of the pathogen or death of any cause | Within 28 days after end of treatment
Number of days admitted related to urinary tract symptoms | Within 28 days after treatment initiation

SECONDARY OUTCOMES:
Number of days with antibiotic-related non-serious adverse events. | From date of treatment initiation until the date of treatment stop for the baseline infection, assessed up to 14 days
  Data on diarrhea, loss of appetite, and vomiting will be included.
Proportion of participants with a recurrent urinary tract infection regardless of the pathogen or death of any cause. | Within 100 days after end of treatment
Proportion of participants with a recurrent infection with a bacterium resistant to the antibiotic given for the baseline infection or an opportunistic infection | Within 100 days after end of treatment

OTHER OUTCOMES:
Proportion of participants with a serious adverse event. | Within 100 days after treatment initiation
  Defined as any untoward medical occurrence that results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in persistent or significant disability, or jeopardizes the patient

CONTACTS AND LOCATIONS:
Overall Officials: Naqash Sethi, MD, Principal Investigator — Department of Pediatrics and Adolescent Medicine, Rigshospitalet, Copenhagen, Denmark; Ulrikka Nygaard, Ass. prof, Ph.D., Study Chair — Department of Pediatrics and Adolescent Medicine, Rigshospitalet, Copenhagen, Denmark
Locations (4):
- Denmark (4):
  - Copenhagen University Hospital Rigshospitalet, Copenhagen
  - Copenhagen University Hospital Herlev, Herlev
  - Copenhagen University Hospital Hillerød, Hillerød
  - Copenhagen University Hospital Hvidovre, Hvidovre

IPD SHARING:
Plan to Share IPD: Yes
Study protocol and statistical analysis plan will be shared. Individual participant data will be shared to facilitate the conduction of research or quality improvement projects.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Primarily for the conduction of research or quality improvement projects.